CLINICAL TRIAL: NCT04455698
Title: Engaging and Activating Cancer Survivors in Genetic Services Study
Acronym: ENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: University of Pennsylvania (Other); St. Jude Children's Research Hospital (Other); Fox Chase Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIRB21-0176; R01CA237369 (NIH)
Record Dates: First submitted 2020-06-25; First posted 2020-07-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remote Telegenetics: TELEPHONE (ARM A) (Experimental): Remote Phone Telegenetics:
  Participants with complete pre-test and disclosure counseling with a Genetic Counselor using remote services - TELEPHONE.
  Interventions: Behavioral: Remote Telegenetic Counseling by Phone
- Remote Telegenetics: VIDEOCONFERENCING (ARM B) (Experimental): Remote Videoconferencing Telegenetics:
  Participants with complete pre-test and disclosure counseling with a Genetic Counselor using remote services - VIDEOCONFERENCING.
  Interventions: Behavioral: Remote Telegenetic Counseling by Videoconferencing
- USUAL CARE (ARM C) (Experimental): Usual Care:
  Participants will receive referrals to genetic counseling providers, initiating services on their own. At 6 months, if participants have not sought and received genetic counseling services, they will be offered randomization to ARM A/ARM B.
  Interventions: Behavioral: Usual Care Arm

INTERVENTIONS:
Behavioral: Remote Telegenetic Counseling by Phone — Participants will receive standard of care pre-test and disclosure genetic counseling with a genetic counselor by Telephone.
  Arms: Remote Telegenetics: TELEPHONE (ARM A)
Behavioral: Remote Telegenetic Counseling by Videoconferencing — Participants will receive standard of care pre-test and disclosure genetic counseling with a genetic counselor using Videoconferencing Technology.
  Arms: Remote Telegenetics: VIDEOCONFERENCING (ARM B)
Behavioral: Usual Care Arm — Participants in the usual care arm will receive usual care services depending on which referral method they choose and if they initiate services. After a 6 month status survey, if they have not had genetic services through usual care they will be offered services and re-randomized to ARM A/ARM B.
  Arms: USUAL CARE (ARM C)

SUMMARY:
To address the gap in access to genetic services, this study will evaluate the effectiveness of an adapted model of remote delivery of genetic services to increase the uptake of recommended genetic assessment and testing in childhood cancer survivors.

DETAILED DESCRIPTION:
As childhood cancer survivors receive care locally from PCPs, the in-home, collaborative PCP model is designed to increase access to genetic services and uptake of genetic testing in childhood cancer survivors. In this model, individual survivors can access remote telegenetic services and genetic counselors will partner with PCPs to order genetic testing.

This study comprises of a 3-arm randomized Hybrid 1 Effectiveness and Implementation study in 360 CCSS survivors to evaluate the effectiveness of our in-home, collaborative PCP model of remote telegenetic services to increase uptake of cancer genetic testing in childhood cancer survivors compared to usual care options for genetic testing.

Aims are as follows:

To evaluate the effectiveness of our in-home, collaborative PCP model of remote telegenetic services to increase uptake of genetic testing at 6 months as compared to usual care among childhood cancer survivors who meet criteria for cancer genetic testing. Our primary outcome will be a composite variable indicating whether a person had pre-test counseling or genetic testing.

To evaluate the effectiveness of remote videoconferencing to provide greater increase in knowledge and decrease in distress and depression as compared to remote phone services, to examine the moderators of patient outcomes with remote telegenetic services, and to estimate intervention costs and incremental cost-effectiveness of the three study arms.

To conduct a multi-stakeholder, mixed-methods process evaluation to understand patient, provider and system factors associated with uptake of counseling and testing in our adapted in-home, collaborative PCP model and facilitators and barriers to uptake to provide recommendations for future implementation.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and communicate in English or Spanish
* Currently residing in the US
* Childhood Cancer Survivor Study Participant survivors of the following primary cancers:

  * CNS tumor
  * Sarcoma (except Ewing sarcoma)
  * Hepatoblastoma
  * Leukemia
* Childhood Cancer Survivor Study Participant with a family history of a child with cancer:

  * 2 or more malignancies in childhood (age 18 or younger)
  * A first degree relative (parent or sibling) with cancer aged 45 or younger
  * 2 or more second degree relatives with cancer aged 45 or younger (same side of family)
  * Parents of the child with cancer are related (consanguinity)
  * Other family history that meets NCCN criteria
* Able to communicate remotely through remote telegenetic platforms (phone or videoconference) with genetic counselors

Exclusion Criteria:

* Uncorrected or uncompensated speech defects that would lead to the participant being unable to communicate effectively with genetic counselor
* Currently residing in a US state or territory where genetic counselors are not licensed to provide care
* Uncontrolled psychiatric/mental condition or severe physical, neurological or cognitive deficits rendering individual unable to understand study goals and task
* Participants who have already completed and received a clinically appropriate multi-gene panel genetic testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who received testing or genetic counseling | 6 Months status survey (ARM C)
  Primary composite outcome collected via remote services records-Yes/No (ARMS A/B)
Genetic Knowledge Scale | Baseline - Within 7 Days After Result Disclosure
  Change in knowledge (ARMS A/B only). Increased change score indicates increase in knowledge (better).
Impact of Events Scale (IES) | Baseline - Within 7 Days After Result Disclosure
  Change in Cancer Specific Distress (ARMS A/B only). Score Range = 0-40. Decreased score change indicates a decrease in distress (better).
Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline - Within 7 Days After Result Disclosure
  Change in Depression (ARMS A/B only). Score Range = 4-20. Decreased score change indicates a decrease in depression (better).

SECONDARY OUTCOMES:
Uptake of genetic counseling, testing, and identification of genetic carriers | 6 month status survey (ARM C)
  Collected via remote services records (ARMS A/B)
Patient Reported Outcomes Measurement Information Systems (PROMIS) | Baseline - Within 7 Days After Result Disclosure
  Change in Anxiety (ARMS A/B only). Score Range = 4-20. Decreased score change indicates a decrease in anxiety (better).
Multi-dimensional Impact of Cancer Risk Assessment Questionnaire (MICRA) | Baseline - Within 7 Days After Result Disclosure
  Change in Uncertainty (ARMS A/B only). Score Range = 0-85. Decreased score change indicates a decrease in uncertainty (better).
Change in Health Behaviors (Selected from the Behavioral Risk Factor Surveillance System Questionnaire and the Health and Diet survey Dietary Guidelines Supplement) | Baseline - 6 Months After Result Disclosure
  Change in performance of risk reductive and screening behaviors and communication of results - Yes/No responses (ARMS A/B only).

CONTACTS AND LOCATIONS:
Overall Officials: Tara O Henderson, MD, MPH, Principal Investigator — University of Chicago; Angela Bradbury, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - St Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henderson TO, Egleston B, Howe S, Allen MA, Mim R, Fleisher LG, Elkin EB, Oeffinger KC, Krull KR, Ofidis D, Mcleod B, Griffin H, Wood EM, Cacioppo CN, Brown S, Perpich M, Armstrong GT, Bradbury AR. The ENGAGE Study: A Randomized Trial Optimizing Uptake of Germline Cancer Genetic Services in Childhood Cancer Survivors. medRxiv [Preprint]. 2025 Oct 22:2025.10.20.25338173. doi: 10.1101/2025.10.20.25338173. PMID 41282828
- [Derived] Henderson TO, Allen MA, Mim R, Egleston B, Fleisher L, Elkin E, Oeffinger K, Krull K, Ofidis D, Mcleod B, Griffin H, Wood E, Cacioppo C, Weinberg M, Brown S, Howe S, McDonald A, Vukadinovich C, Alston S, Rinehart D, Armstrong GT, Bradbury AR. The ENGAGE study: a 3-arm randomized hybrid type 1 effectiveness and implementation study of an in-home, collaborative PCP model of remote telegenetic services to increase uptake of cancer genetic services in childhood cancer survivors. BMC Health Serv Res. 2024 Feb 28;24(1):253. doi: 10.1186/s12913-024-10586-z. PMID 38414045

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT04455698/Prot_SAP_ICF_000.pdf